CLINICAL TRIAL: NCT06906770
Title: Virtual Reality-based Eye Movement Desensitisation and Reprocessing Therapy for Specific Phobias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Northampton (Other)
Collaborators: St Andrew's Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHSHEA000372
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Specific Phobias
Keywords: Eye Movement Desensitization and Reprocessing (EMDR); Virtual Reality
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR EMDR (Experimental)
  Interventions: Other: Eye movement desensitization and reprocessing phobia treatment in virtual reality

INTERVENTIONS:
Other: Eye movement desensitization and reprocessing phobia treatment in virtual reality — Short form and frequent eye movement desensitization and reprocessing (EMDR) in virtual reality for specific phobia treatment.

SUMMARY:
The goal of this clinical trial is to study the effectiveness of a virtual reality-based eye movement desensitization and reprocessing (EMDR) application in treating phobia. It will also learn about the feasibility and safety of the application for independent use.

The main questions it aims to answer are:

Does the VR EMDR application reduce distress, improve positive cognitions, and decrease avoidance of specific phobias? Can the application help diminish phobia-related bodily sensations and encourage cognitive shifts toward positive beliefs and greater confidence in confronting previously avoided situations? Can the participants independently administer the treatment with minimum assistance?

Participants will:

Visit the site and take the VR EMDR phobia treatment every day for one week. Report their phobia and simulator sickness symptoms through self-report questionnaires or semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Have a specific phobia (not necessarily clinically significant)

Exclusion Criteria:

* Diagnosis of mental health disorders
* History of trauma associated with their phobia
* History of panic attacks associated with their phobia
* History of psychosis
* Current self-harm
* Current suicidal ideation
* Regular use of substances that might affect mental state
* Regular use of medications that might affect mental state
* Significant visual impairments
* Severe motion sickness

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Units of Distress (SUDs) | Recorded 4 times during each VR EMDR session (first being baseline, and the subsequent three were recorded after each eye movement set in desensitisation phrase) across the 5 consecutive intervention days.
  The Subjective Units of Distress Scale (SUDs) is a self-reported measure of distress experienced by participants during each virtual reality (VR) EMDR session. Participants will rate their level of distress on a scale from 0 (no distress) to 10 (highest distress). Outcome is measured by the change in SUD score throughout each session and cumulative change from Day 1 to Day 5.
Change in Validity of Cognitions (VoC) | Recorded 4 times during each VR EMDR session (first being baseline, and the subsequent three were recorded after each eye movement set in installation phrase) across the 5 consecutive intervention days.
  The Validity of Cognition (VoC) scale measures the strength of positive cognitions related to the phobic trigger. Participants will rate how true their preferred positive cognition feels on a scale from 1 (completely false) to 7 (completely true) during each VR EMDR session. Outcome is measured by change in VoC score throughout each session and cumulative change from Day 1 to Day 5.
Change in IAPT Phobia Scale Score | Baseline (Day 0, pre-intervention) and post-intervention (Day 5).
  The Improving Access to Psychological Therapies (IAPT) Phobia Scale assesses the severity of phobic symptoms in terms of avoidance behaviour. Participants will complete the scale before the intervention (baseline) and immediately after the final session (Day 5). Outcome is measured by the change in IAPT Phobia Scale score from baseline to Day 5 post-intervention. Participants achieved remission if they scored below the threshold of 4 in the Improving Access to Psychological Therapies Phobia (IAPT) phobia scale.
The Severity Measure for Specific Phobia-Adult | Baseline (Day 0, pre-intervention) and post-intervention (Day 5).
  The Severity Measure for Specific Phobia-Adult is a 10-item measure that assesses the severity of specific phobia in individuals age 18 and older. The measure was designed to be completed by an individual upon receiving a diagnosis of specific phobia (or clinically significant specific phobia symptoms) and thereafter, prior to follow-up visits with the clinician. Each item asks the individual to rate the severity of his or her specific phobia during the past 7 days.

SECONDARY OUTCOMES:
Simulator Sickness Questionnaire (SSQ) Score Change | Day 1 and Day 5 post-intervention.
  The Simulator Sickness Questionnaire (SSQ) is used to assess potential side effects of virtual reality exposure, including nausea, oculomotor discomfort, and disorientation. Participants will complete the SSQ at the end of the first and last intervention days. Outcome is measured by the change in total SSQ score between Day 1 and Day 5.
Participant Adherence | Day 5 post-intervention.
  Description: Adherence will be assessed based on the number of sessions completed
Participant Acceptability | Day 5 post-intervention
  Description: Acceptability will be evaluated using participant feedback collected at the end of the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Northampton, Northampton, Northamptonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The increased risk of patients being identified.